CLINICAL TRIAL: NCT02920580
Title: The NEUROlogically-impaired Extubation Timing Trial
Acronym: NEURO-ETT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Damon Scales, MD, PhD, FRCPC, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NEURO-ETT (Vanguard)
Record Dates: First submitted 2016-09-22; First posted 2016-09-30 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Acute Brain Injury
Keywords: Subarachnoid hemorrhage; Spontaneous intracerebral hemorrhage; Global cerebral anoxia/cardiac arrest; Meningitis/Encephalitis/Cerebral abscess; Seizure; Traumatic Brain Injury (TBI); Ischemic Stroke; Brain tumor
MeSH Terms: conditions — Brain Injuries; Subarachnoid Hemorrhage; Heart Arrest; Meningitis; Seizures; Brain Injuries, Traumatic; Ischemic Stroke; Brain Neoplasms | interventions — Airway Extubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extubation (Active Comparator): Extubation by removal of endotracheal tube.
  Interventions: Procedure: Extubation
- Usual care (Active Comparator): The usual clinical practice is removal of the endotracheal tube (extubation), or insertion of tracheostomy, timed according to physicians' discretion
  Interventions: Procedure: Usual Care

INTERVENTIONS:
Procedure: Extubation — This is an extubation by removal of endotracheal tube which must be done on the day of randomization or the following day. Any decision to subsequently reintubate the patient will be left to the discretion of the clinical team. Similarly, if a tracheostomy is deemed necessary in a patient who fails the extubation attempt, this will be managed at the discretion of the treating team. If for any reason the patient is not extubated according to the randomized schedule, the reason(s) will be recorded on a protocol violation form and the site investigator will be notified. If a patient receives a tracheostomy instead of being extubated we will again record reasons for this, but the patient will be analysed in the extubation group according to the intention-to-treat principle.
  Arms: Extubation
Procedure: Usual Care — Patients in this group will be treated according to usual care, which may include extubation (removal of endotracheal tube) or insertion of a tracheostomy, timed according to physicians' discretion. The inclusion of this arm will allow prompt extubation to be compared to usual practice, which often involves further observation and delayed decision-making due to clinician uncertainty about the optimal airway management strategy. Incorporation of usual care arms has been promoted as a design feature to improve the safety and interpretability of critical care clinical trials.
  Arms: Usual care

SUMMARY:
This randomized controlled trial will enrol patients with acute severe brain injury who pass a spontaneous breathing trial but have decreased level of consciousness. It will directly compare (1) prompt extubation vs. (2) usual care, with extubation or tracheostomy timed according to physicians' discretion. The primary outcome will be ICU free days (days spent alive and outside an ICU).

DETAILED DESCRIPTION:
Thousands of patients suffer severe brain injuries every year, from causes such as trauma, stroke, and infection. Extensive clinical research in weaning from mechanical ventilation has led to recommendations for prompt extubation following a successful trial of spontaneous breathing in general intensive care unit (ICU). However, little evidence exists to guide decisions about when to remove the breathing tube in patients with severe brain injury. It is unclear which of the following strategies would optimize important patient outcomes: prompt extubation vs. waiting and extubating or performing a tracheostomy, timed according to physicians' discretion. Each strategy has associated risks: prompt extubation may lead to higher rates of extubation failure and reintubation, whereas waiting longer may expose patients to complications from prolonged mechanical ventilation and tracheostomy may lead to procedural complications (or unnecessary procedures, if prompt extubation would be successful). This trial in brain-injured patients will test which of the following will lead to better patient outcomes: (1) removing the endotracheal tube promptly once a spontaneous breathing trial is passed; or (2) usual care, with the airway management strategy selected according to the preference of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years
* Acute brain injury (subarachnoid hemorrhage, ischemic stroke, spontaneous intracerebral hemorrhage, seizure, traumatic brain injury, brain tumor, global cerebral anoxia/cardiac arrest, meningitis/encephalitis/cerebral abscess) that occurred within the previous 4 weeks.
* Receiving invasive mechanical ventilation via endotracheal tube for > 72 hours
* Glasgow Coma Scale motor score 3 to 6 with improvement or no change from previous day
* passed spontaneous breathing trial (SBT)

Exclusion Criteria:

* Previous extubation during this ICU admission
* Quadriplegic
* Neuromuscular disease that will result in prolong need for mechanical ventilation, including but not limited to Guillain-Barre syndrome, cervical spinal cord injury, advanced multiple sclerosis
* Do-Not-Reintubate order in place
* Previously randomized in this trial
* Underlying pre-existing condition with expected mortality less than 6-months.
* Anticipated/scheduled for surgical procedures within 48 hours
* C-spine not yet cleared for activity as tolerated (cleared for activity as tolerated while wearing hard collar is acceptable)
* Currently known or suspected to have an difficult airway
* Absence of an endotracheal tube cuff leak, if checked
* Absence of spontaneous or induced cough
* Current enrolment in an RCT that precludes NEURO-ETT co-enrollment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
ICU Free Days | 60 days
  The primary outcome is number of ICU free days to day 60, defined as the number of days spent alive and outside of an ICU until day 60.
  The primary outcome will be measured to answer the following primary question: Among patients receiving minimal mechanical ventilatory support for severe and persistent brain injury, which of the following airway management strategies increase ICU-free days to day 60: (1) prompt extubation vs. (2) usual care, which may include extubation or tracheostomy timed according to physicians' discretion?

SECONDARY OUTCOMES:
Mortality, | up to 6 months
  Mortality at ICU discharge, mortality at hospital discharge, mortality at 3 months, mortality at 6 months
Ventilator-Free Days | up to 60 days
  Days free of mechanical ventilation, total duration (days) of ventilation among survivors
Airway Complications | up to 60 days
  Presence versus absence of airway complication
Nutrition Intake | up to 6 months
  Time to normal oral nutrition intake
Antibiotic Days | up to day 14
  Injection or infusion of antibiotics given intravenously
Delirium | up to day 14
  Presence versus absence of delirium experienced
Rate of Tracheostomy Insertion | up to 6 months
  Presence versus absence of tracheostomy insertion
Rate of ICU Readmission | up to hospital discharge
  ICU readmission rates to hospital discharge
Hospital Discharge Destination | at hospital discharge
  Destination of the patient post hospitalization - home, rehabilitation facility, retirement home, long-term care/nursing home, no fixed address or shelter, continuing complex care, acute care hospital, other
Extended Glasgow Outcome Score | up to 6 months
  Functional outcome (scoring 1 to 8)
EQ-5D | up to 6 months
  Health related quality of life (scoring 1 to 5)

CONTACTS AND LOCATIONS:
Overall Officials: Niall Ferguson, MD, MSc,, Principal Investigator — Toronto General Hospital; Damon Scales, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (13):
- Canada (13):
  - University of Alberta Hospital, Edmonton, Alberta
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - L'Hôpital de l'Enfant-Jésus, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No